CLINICAL TRIAL: NCT02427802
Title: A Phase 3 Randomized, Placebo-Controlled, Blinded Study to Investigate the Safety and Efficacy of a Topical Gentamicin-Collagen Sponge in Combination With Systemic Antibiotic Therapy in Diabetic Patients With an Infected Foot Ulcer
Brief Title: Study of a Topical Gentamicin-Collagen Sponge Along With Systemic Antibiotic in Infected Diabetic Foot Ulcers
Acronym: COACT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INN-TOP-004
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Foot Ulcer, Diabetic; Infection
MeSH Terms: conditions — Diabetic Foot; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gentamicin sponge group (Experimental): Topical Gentamicin Collagen Sponge: Up to four collagen sponges each containing 50 mg of gentamicin sulfate (equivalent to 32.5 mg of gentamicin base) administered daily, with systemic antibiotic therapy and standard ulcer care (gentamicin-sponge group) for up to 28 days.
  Interventions: Drug: Gentamicin collagen sponge
- Placebo sponge group (Placebo Comparator): Matching placebo collagen sponge administered daily, with systemic antibiotic therapy and standard ulcer care (gentamicin-sponge group) for up to 28 days.
  Interventions: Other: Placebo
- No sponge group (No Intervention): Systemic antibiotic therapy and standard ulcer care (gentamicin-sponge group) for up to 28 days.

INTERVENTIONS:
Drug: Gentamicin collagen sponge — Up to 4 topical Gentamicin Collagen Sponges each containing 50 mg of gentamicin sulfate (equivalent to 32.5 mg of gentamicin base)
  Other Names: Cogenzia
  Arms: Gentamicin sponge group
Other: Placebo — Matching collagen sponge
  Arms: Placebo sponge group

SUMMARY:
This is a phase 3, randomized, controlled, blinded, multicenter study conducted in 3 parallel cohorts of diabetic patients with at least 1 infected foot ulcer. Patients will be randomized to receive 1 of 3 study treatments; systemic antibiotic therapy and standard ulcer care with either (A) daily application of a gentamicin-sponge, (B) daily application of a placebo-sponge or (C) no-sponge, in the ratio 2:1:1.

Patients will be treated for approximately 28 days and return to the clinic weekly for safety and efficacy assessments. After completing treatment, patients will return to the clinic for scheduled follow-up visits approximately 10, 30, 60 and 90 days after treatment is stopped.

DETAILED DESCRIPTION:
This is a phase 3, randomized, controlled, blinded, multicenter study conducted in 3 parallel cohorts of diabetic patients with at least 1 infected foot ulcer. Patients will be randomized using an electronic randomization system to receive 1 of 3 study treatments; systemic antibiotic therapy and standard ulcer care with either (A) daily application of a gentamicin-sponge, (B) daily application of a placebo-sponge or (C) no-sponge, in the ratio 2:1:1. The investigator will be blinded to the patient's treatment group assignment and patients randomized to one of the 2 sponge groups will be blinded as to whether the sponge is active or placebo.

If a patient has multiple infected ulcers, the assigned treatment will be administered to all infected ulcers. The investigator will determine the highest severity ulcer to be used for all efficacy evaluations and will also determine the size and number of sponges (up to 4) that a patient will use in order to completely cover all infected ulcers. The investigator will prescribe an empiric systemic antibiotic therapy based on protocol instructions.

Patients will be treated for approximately 28 days and return to the clinic weekly for safety and efficacy assessments. The investigator will stop study treatment if a patient achieves clinical cure by or after the 3rd treatment visit (approximately study day 15). After completing treatment, patients will return to the clinic for scheduled follow-up visits or until ulcer closure. The final efficacy assessments used in the primary efficacy analyses will be obtained at the first follow-up visit approximately 10 days after treatment is stopped. The remaining follow-up visits will occur at approximately 30, 60 and 90 days after treatment is stopped when patients will be assessed for ulcer closure and any re-infection.

ELIGIBILITY:
Inclusion Criteria:

* Has diabetes mellitus, according to the American Diabetes Association (ADA) criteria.
* Has at least 1 skin ulcer located on or below the malleolus that presents with the following clinical manifestations of a moderate or severe infection based on the Infectious Disease Society of America guidelines for the "Diagnosis and Treatment of Diabetic Foot Infections" (CID 2012; 54:132-173) (IDSA guidelines):

  * has ≥ 2 manifestations of inflammation (local swelling or induration, erythema, local tenderness or pain, local warmth, purulent discharge (thick, opaque to white or sanguineous secretion)
  * has ≥ 1 of the following characteristics: erythema > 2cm, or involving structures deeper than skin and subcutaneous tissues (e.g. abscess, osteomyelitis, septic arthritis, fasciitis) For patients with multiple infected ulcers, the ulcer with the highest Diabetic Foot Infection Wound score (DFI score) must be on or below the malleolus and all infected ulcers must be completely coverable using no more than 4 sponges (sponges cannot be cut).
* Has documented adequate arterial perfusion in the affected limb(s) (either palpable dorsalis pedis and posterior tibial pulses, or normal Doppler wave forms, a toe blood pressure ≥ 45 mm Hg or participation is approved by a vascular surgeon)
* Has received appropriate surgical intervention to remove all necrotic and infected bone if diagnosed with osteomyelitis.
* Has received appropriate surgical debridement to remove all gangrenous tissue.

Exclusion Criteria:

* Has a known history of hypersensitivity to gentamicin (or other aminoglycosides).
* Has a known or suspected hypersensitivity to bovine collagen.
* Has an ulcer infection which, based upon the patient's known history of hypersensitivity and/or as otherwise in the opinion of the investigator, cannot be adequately treated with at least one of the empiric systemic antibiotic regimens allowed by this protocol.
* Has an ulcer associated with prosthetic material or an implanted device.
* Has received any systemic or topical antibiotic therapy for any reason within 7 days of randomization unless it was administered to specifically treat the infected ulcer(s) and only within 36 hours of randomization.
* Requires or is likely to require treatment with any concomitant topical product or wound therapy before the first follow-up study visit.
* Is severely immunocompromised, or likely to become severely immunocompromised during the study, in the opinion of the investigator.
* Has a history of myasthenia gravis or other neurological condition where gentamicin use is contraindicated as determined by the investigator.
* Has a history of epilepsy.
* Has a history of alcohol or substance abuse in the past 12 months.
* Has an uncontrolled illness that, in the opinion of the investigator, is likely to cause the patient to be withdrawn from the trial or would otherwise interfere with interpreting the results of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Jones, Study Director — Vice President, Global Clinical Operations, Innocoll Pharmaceutical
Locations (70):
- United States (70):
  - Anniston, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chino, California
  - Corona, California
  - Fountain Valley, California
  - Fresno, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - San Francisco, California
  - Sylmar, California
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Clermont, Florida
  - Cooper City, Florida
  - Coral Gables, Florida
  - DeLand, Florida
  - Fleming Island, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Miami Springs, Florida
  - New Port Richey, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Weston, Florida
  - Augusta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Idaho Falls, Idaho
  - Avon, Indiana
  - Mooresville, Indiana
  - Muncie, Indiana
  - Baltimore, Maryland
  - Phoenix, Maryland
  - Boston, Massachusetts
  - Flint, Michigan
  - Butte, Montana
  - Great Falls, Montana
  - Las Vegas, Nevada
  - North Brunswick, New Jersey
  - Somerset, New Jersey
  - Hopewell Junction, New York
  - New Windsor, New York
  - Durham, North Carolina
  - Lima, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - West Columbia, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Lampasas, Texas
  - Lubbock, Texas
  - McAllen, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Webster, Texas
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Started | 305 | 154 | 153
Completed | 246 | 120 | 110
Not Completed | 59 | 34 | 43
Not completed — Adverse Event | 11 | 3 | 7
Not completed — Death | 0 | 4 | 1
Not completed — Lost to Follow-up | 13 | 8 | 8
Not completed — Physician Decision | 4 | 2 | 4
Not completed — Withdrawal by Subject | 10 | 5 | 11
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — protocol specific treatment unrelated | 18 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group | Total
Number analyzed (Participants) | 305 | 154 | 153 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.84) | 57.1 (11.12) | 56.7 (11.16) | 57.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 47 | 34 | 146
  Male | 240 | 107 | 119 | 466
Region of Enrollment [Number; unit: participants]
  United States | 305 | 154 | 153 | 612

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure (Resolution of All Clinical Signs and Symptoms of Infection)
Description: The primary efficacy variable is the percent of patients with a clinical outcome of clinical cure (Resolution of all clinical signs and symptoms of infection) at F/U visit 1
Time Frame: approximately 10 days after end of treatment
Population: modified intent to treat population consisted of randomized patients who received any dose of gentamicin-sponge or placebo-sponge or who were randomized to the no sponge arm, and who were not early-terminated for any of the treatment-unrelated reasons before F/U visit 1,
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 283 | 141 | 140
Participants | 115 | 64 | 48

2. Secondary Outcome: Clinical Cure and Baseline Pathogen Eradication (Resolution of All Clinical Signs and Symptoms of Infection) and Baseline Pathogen Eradication)
Description: Percent of patients with both a clinical outcome of clinical cure (Resolution of all clinical signs and symptoms of infection) and baseline pathogen eradication at F/U visit 1
Time Frame: Approximately 10 days after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 283 | 141 | 140
Participants | 87 | 47 | 34

3. Secondary Outcome: Reinfection (Percent of Patients With Re-infection)
Description: Percent of patients with re-infection
Time Frame: Approximately 90 days after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 283 | 141 | 140
Participants | 12 | 5 | 2

4. Secondary Outcome: Time to Clinical Cure
Description: Actual time to clinical cure (Resolution of all clinical signs and symptoms of infection)
Time Frame: Approximately 10 days after end of treatment
Population: Modified Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 140 | 75 | 59
Days | 41 [30.0 to NA] — Upper boundary not reached | 33 [29.0 to NA] — Upper boundary not reached | 46 [30.0 to NA] — Upper boundary not reached

5. Secondary Outcome: Amputation (Percent of Patients That Have an Amputation Associated With the Target Ulcer)
Description: Percent of patients that have an amputation associated with the target ulcer
Time Frame: Within approximately 90 days of end of treatment
Population: Modified Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 283 | 141 | 140
Participants | 2 | 3 | 5

6. Secondary Outcome: Ulcer Closure (Percent of Patients With Target Ulcer Closure)
Description: Percent of patients with ulcer closure within approximately 30 days of end of treatment
Time Frame: within approximately 30 days of end of treatment
Population: Modified Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
Number analyzed (Participants) | 283 | 141 | 140
Participants | 67 | 32 | 29

ADVERSE EVENTS:
Time Frame: approximately 28 days
Arm/Group | Gentamicin Sponge Group | Placebo Sponge Group | No Sponge Group
All-Cause Mortality (participants affected / at risk) | 0/305 | 4/154 | 1/153
Serious Adverse Events (participants affected / at risk) | 44/305 | 22/154 | 26/153
Other Adverse Events (participants affected / at risk) | 135/305 | 72/154 | 65/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sponge Group (N=305) | Placebo Sponge Group (N=154) | No Sponge Group (N=153)
osteomyelitis (Infections and infestations) | 7 (7) | 4 (4) | 7 (7)
infected skin ulcer (Infections and infestations) | 7 (7) | 1 (1) | 4 (4)
cellulitis (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
osteomyelitis acute (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
gangrene (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
cardiac failure congestive (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
diabetes mellitus inadequate cotnrol (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
pulmonay embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
death (General disorders) | 0 (0) | 0 (0) | 1 (1)
device extrusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
hip fracture (General disorders) | 1 (1) | 0 (0) | 0 (0)
limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
penile necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sponge Group (N=305) | Placebo Sponge Group (N=154) | No Sponge Group (N=153)
infected skin ulcer (Infections and infestations) | 23 (23) | 11 (11) | 8 (8)
Osteomyelitis (Infections and infestations) | 10 (10) | 8 (8) | 10 (10)
Cellulitis (Infections and infestations) | 7 (7) | 4 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Sepsis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Upper Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 22 (22) | 13 (13) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
skin ulcer (Skin and subcutaneous tissue disorders) | 26 (26) | 9 (9) | 11 (11)
Blister (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 0 (0)
Type 2 diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 7 (7) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (4)
Acute Kidney Injury (Renal and urinary disorders) | 8 (8) | 4 (4) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 12 (12) | 4 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 3 (3) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of the multicenter study had to be published prior to the publication of any site specific data.